CLINICAL TRIAL: NCT02140255
Title: Very Early Intensive Treatment of Infants Living With HIV to Achieve HIV Remission: A Phase I/II Proof of Concept Study
Brief Title: Very Early Intensive Treatment of Infants Living With HIV to Achieve HIV Remission
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT P1115; UM1AI068632 (NIH); UM1AI068616 (NIH); UM1AI106716 (NIH); 11954 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-04

CONDITIONS: HIV Infection
Keywords: HIV Remission
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Lopinavir; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1, Regimen 1L: 2 NRTIs + NVP + LPV/r (Experimental): Participants will receive 2 NRTIs + NVP + LPV/r.
  Interventions: Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs); Drug: Nevirapine (NVP); Drug: Lopinavir/Ritonavir (LPV/r)
- Cohort 2, Regimen 1L: 2 NRTIs + NVP + LPV/r (Experimental): Participants will receive 2 NRTIs + NVP + LPV/r.
  Interventions: Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs); Drug: Nevirapine (NVP); Drug: Lopinavir/Ritonavir (LPV/r)
- Cohort 1, Regimen 2R: 2 NRTIs + NVP + RAL (Experimental): Participants will receive 2 NRTIs + NVP + RAL.
  Interventions: Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs); Drug: Nevirapine (NVP); Drug: Raltegravir (RAL)
- Cohort 2, Regimen 2R: 2 NRTIs + NVP + RAL (Experimental): Participants will receive 2 NRTIs + NVP + RAL.
  Interventions: Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs); Drug: Nevirapine (NVP); Drug: Raltegravir (RAL)
- Cohort 1, Regimen 2RV: 2 NRTIs + NVP + RAL + VRC01 (Experimental): Participants will receive 2 NRTIs + NVP + RAL + VRC01.
  Interventions: Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs); Drug: Nevirapine (NVP); Drug: Raltegravir (RAL); Drug: VRC01
- Cohort 1, Regimen 3RD: 2 NRTIs + NVP + RAL switch to 2 NRTIs + DTG (Experimental): Participants will receive 2 NRTIs + NVP + RAL with subsequent switch to 2 NRTIs + DTG upon reaching 28 days of age and 3 kg body weight.
  Interventions: Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs); Drug: Nevirapine (NVP); Drug: Raltegravir (RAL); Drug: DTG
- Cohort 1, Regimen 3RDV7: 2 NRTIs + NVP + RAL + VRC07-523LS switch to 2 NRTIs + DTG + VRC07-523LS (Experimental): Participants will receive 2 NRTIs + NVP + RAL + VRC07-523LS with subsequent switch to 2 NRTIs + DTG + VRC07-523LS upon reaching 28 days of age and 3 kg body weight.
  Interventions: Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs); Drug: Nevirapine (NVP); Drug: Raltegravir (RAL); Drug: VRC07-523LS

INTERVENTIONS:
Drug: Nucleoside Reverse Transcriptase Inhibitors (NRTIs) — Chosen by the site investigator and dosed according to World Health Organization (WHO) or individual country or local standard guidelines.
Drug: Nevirapine (NVP) — Administered orally. Dosed according to study step/participant's age/participant's weight.
Drug: Lopinavir/Ritonavir (LPV/r) — Administered orally. Dosed according to study step and participant's age.
  Arms: Cohort 1, Regimen 1L: 2 NRTIs + NVP + LPV/r; Cohort 2, Regimen 1L: 2 NRTIs + NVP + LPV/r
Drug: Raltegravir (RAL) — Administered orally. Dosed according to study step and participant's age.
  Arms: Cohort 1, Regimen 2R: 2 NRTIs + NVP + RAL; Cohort 1, Regimen 2RV: 2 NRTIs + NVP + RAL + VRC01; Cohort 1, Regimen 3RD: 2 NRTIs + NVP + RAL switch to 2 NRTIs + DTG; Cohort 1, Regimen 3RDV7: 2 NRTIs + NVP + RAL + VRC07-523LS switch to 2 NRTIs + DTG + VRC07-523LS; Cohort 2, Regimen 2R: 2 NRTIs + NVP + RAL
Drug: VRC01 — 40 mg/kg administered subcutaneously.
  Arms: Cohort 1, Regimen 2RV: 2 NRTIs + NVP + RAL + VRC01
Drug: DTG — Administered orally. Dosed according to participant's weight.
  Arms: Cohort 1, Regimen 3RD: 2 NRTIs + NVP + RAL switch to 2 NRTIs + DTG
Drug: VRC07-523LS — 40 mg/kg administered subcutaneously.
  Arms: Cohort 1, Regimen 3RDV7: 2 NRTIs + NVP + RAL + VRC07-523LS switch to 2 NRTIs + DTG + VRC07-523LS

SUMMARY:
The study will explore the effects of early intensive antiretroviral therapy (ART) with or without a broadly neutralizing antibody (bNAb) on achieving HIV remission (HIV RNA below the limit of detection of the assay) among infants living with HIV.

DETAILED DESCRIPTION:
The purpose of this study is to explore the effects of early intensive antiretroviral therapy (ART) on achieving HIV remission (HIV RNA below the limit of detection of the assay) among infants living with HIV.

The study will enroll two cohorts. Cohort 1 will include infants born to a mother with presumed or confirmed HIV infection who received no or very limited antiretrovirals during pregnancy. Cohort 2 will include infants with at least one positive HIV nucleic acid test result from a sample collected within 48 hours of birth who initiated a qualifying ART regimen within 48 hours of birth.

Five early intensive therapy regimens will be assessed. Regimen 1L will include 2 nucleoside reverse transcriptase inhibitors (NRTIs) plus nevirapine (NVP) plus lopinavir/ritonavir (LPV/r). Regimen 2R will include 2 NRTIs plus NVP plus raltegravir (RAL). Regimen 2RV will include 2 NRTIs plus NVP plus RAL plus VRC01 monoclonal antibody. Regimen 3RD will include 2 NRTIs plus NVP plus RAL with subsequent switch to 2 NRTIs plus dolutegravir (DTG) upon reaching 28 days of age and 3 kg body weight. Regimen 3RDV7 will include 2 NRTIs plus NVP plus RAL plus VRC07-523LS with subsequent switch to 2 NRTIs plus DTG plus VRC07-523LS upon reaching 28 days of age and 3 kg body weight.

The study will be conducted in four steps. In Step 1, Cohort 1 infants will be enrolled for evaluation of HIV infection and initiation of early intensive therapy within 48 hours of birth. Infants in whom in utero HIV infection is excluded will switch from the study regimen to standard perinatal prophylaxis per local guidelines within two weeks; these infants will continue in Step 1 safety monitoring for two additional weeks, undergo final HIV testing at approximately 24 weeks of age, and then exit the study. Infants in whom in utero HIV infection is confirmed will enter Step 2 at least two weeks after enrollment in Step 1.

In Step 2, infants will receive the study regimen for up to 192 weeks. Beginning at Step 2 Week 84, children who achieved HIV RNA suppression by Week 24, and maintained suppression, thereafter, will be evaluated for possible analytic treatment interruption (ATI).

In Step 3, children in Step 2 who meet criteria for ATI will interrupt ART and be closely monitored for viral rebound for up to five years.

In Step 4, children who experience viral rebound in Step 3 or meet other Step 4 inclusion criteria will re-initiate ART and be closely monitored for viral re-suppression on ART until five years of age or six months after re-suppression, whichever is later.

ELIGIBILITY:
Maternal Inclusion Criteria

1. Presumed or confirmed maternal HIV infection:

   * Mothers will be eligible to enroll with EITHER:

     * Presumed HIV infection defined as at least one positive rapid HIV antibody-based test result from a sample collected in the peripartum period. Presumed infection must be confirmed within 10 business days of enrollment OR
     * Confirmed HIV infection defined as positive results from two samples collected at different timepoints
2. Willing and able to provide written informed consent for participation of herself and her infant. The mother must be of legal age or circumstance to provide independent informed consent as determined by site standard operating procedures (SOPs) and consistent with IRB/EC policies and procedures. Otherwise, informed consent must be obtained from a legal guardian and the mother must provide written assent.
3. Was not previously enrolled in this study with another infant.
4. Did not receive ARVs during the current pregnancy.
5. Infant is eligible per inclusion criteria.

Infant Inclusion Criteria for Step 1

1. Less than or equal to 48 hours of age.
2. Greater than or equal to 36 weeks gestational age at birth (assessment of gestational age will be based on the best clinical estimate determined by date of last menstrual period, antenatal ultrasound, fundal height, or Ballard Score).
3. Greater than or equal to 2 kilograms (kg) at birth.
4. Able to take ARVs by mouth, nasogastric tube, or gastrostomy tube.
5. Has no clinically significant diseases (other than HIV infection) or clinically significant findings during review of medical history or physical examination prior to entry that, in the site investigator's opinion, would interfere with study participation or interpretation.
6. Mother is eligible per inclusion criteria.

Infant Inclusion Criteria for Step 2

1. Enrolled in Step 1.
2. Confirmed in utero HIV infection.
3. Able to take ARVs by mouth, nasogastric tube, or gastrostomy tube.
4. Has no clinically significant diseases (other than HIV infection) or clinically significant findings during review of medical history or physical examination prior to entry that, in the site investigator's opinion, would interfere with study participation or interpretation.
5. Mother (or legal guardian if applicable) is willing and able to provide written informed consent for child's participation in Step 2.

Infant Inclusion Criteria for Step 3

1. Enrolled in Step 2.
2. Has reached Step 2 Week 96.
3. Has the following results based on testing:

   * No confirmed plasma HIV RNA ≥200 copies/mL at Step 2 Week 24 and up to but excluding Step 2 Week 48.
   * No plasma HIV RNA detected at Step 2 Week 48 and thereafter, with two possible exceptions

     * (i) First possible exception: If HIV RNA is detected at or after Step 2 Week 48 with a result <200 copies/mL, testing will be repeated within three weeks (specimen collection for the confirmatory test must occur within three weeks of specimen collection for the initial test).
     * If no HIV RNA is detected on the confirmatory test, or if HIV RNA is detected with a result <200 copies/mL, the infant will be potentially eligible for Step 3 after an additional 48 weeks of follow-up in Step 2, provided no HIV RNA is detected on any subsequent tests in Step 2.
     * If HIV RNA is detected on the confirmatory test with a result ≥200 copies/mL, the infant will not be eligible for Step 3.
     * (ii) Second possible exception: If HIV RNA is detected after Step 2 Week 48 with a result <LOD, the infant will be potentially eligible for Step 3 after an additional 48 weeks of follow-up in Step 2 with no RNA detected. There is no limit on the number of times HIV RNA may be detected with a result <LOD after Week 48. However, infants with detectable RNA with a result <LOD after Week 48 will not be considered for entry into Step 3 until after an additional 48 weeks of no RNA detected.
     * Participants may experience either or both exceptions at different timepoints during follow-up in Step 2.
4. If breastfed, must have permanently ceased breastfeeding, with no exposure to breast milk for at least six weeks prior to specimen collection for the testing specified in the criterion (#5) below.
5. Has met ALL of the following additional criteria while in Step 2, based on testing between Step 2 Week 84 and Step 2 Week 192 (inclusive):

   * Two consecutive negative HIV antibody tests by fourth generation ELISA at least eight weeks apart.
   * Two consecutive HIV DNA tests with no DNA detected in at least 850,000 PBMCs assayed at least eight weeks apart.
   * CD4 cell percentage greater than or equal to 25% and CD4 cell absolute count greater than or equal to the lower limit of normal for age (≥1000 cells/mL if 2 to less than 3 years of age; ≥750 cells/mL if 3 to less than 5 years of age; ≥500 cells/mL if 5 years of age or older).
   * Infant assessed by the site investigator or designee as expected to adhere to the Step 3 Schedule of Evaluations.
   * Mother (or legal guardian if applicable) willing and able to provide written informed consent for child's participation in Step 3 and Step 4.
6. No plasma HIV RNA detected by testing after criteria have been confirmed, with specimen collection for the assay within 14 days prior to Step 3 Entry.

Infant Inclusion Criteria for Step 4

1. Enrolled in Step 3.
2. Has met at least one of the following:

   * Plasma HIV RNA ≥LOD based on two assays.
   * Plasma HIV RNA ≥1000 copies/mL in the presence of fever or other sign or symptom of acute retroviral syndrome.
   * Confirmed or suspected diagnosis of acute retroviral syndrome.
   * Confirmed or suspected diagnosis of a new WHO Clinical Stage 3 or 4 condition.
   * Confirmed CD4 cell percentage less than 25% and CD4 cell absolute count less than the lower limit of normal for age (<1000 cells/mL if 2 to less than 3 years of age; <750 cells/mL if 3 to less than 5 years of age; <500 cells/mL if 5 years of age or older).
   * Otherwise assessed by the site investigator or designee, in consultation with the Clinical Management Committee (CMC), as having an indication to re-initiate treatment.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1120 (Estimated)
Dates: Start 2015-01-23 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve HIV remission | Measured through Week 48
  Defined as no confirmed HIV RNA greater than or equal to the limit of detection (LOD) through 48 weeks of treatment interruption

SECONDARY OUTCOMES:
Frequency of Grade 3 or higher adverse events possibly, probably or definitely related to any component of the study regimen | Measured through Week 192
  Graded according to the DAIDS AE Grading Table, Corrected Version 2.1, dated July 2017
Number of participants with viral suppression to consistent HIV-1 RNA less than LOD | Measured through Week 24
  Based on laboratory evaluations
Number of participants meeting all eligibility criteria for treatment interruption | Measured through Week 192
  As defined in criteria described in study protocol
Number of infants meeting the selected eligibility criteria for treatment interruption among infants who also met the viral suppression criteria for treatment interruption. | Measured through Week 192
  As defined in criteria described in the study protocol
Number of participants who experience HIV persistence | Measured through Week 48
  As measured by plasma viremia (single copy), droplet digital DNA, replication competent HIV reservoirs

OTHER OUTCOMES:
Change in HIV-specific immune response | Measured through Week 48
  As measured by %CD8+/DR+ T cells
Change in immune activation markers (%CD8+/DR+ T cells) response | Measured through Week 48
  As measured by HIV-specific antibodies and HIV-specific T cell responses
Change in DTG concentration among treated neonates and young infants | Measured through Week 24
  Based on laboratory evaluations
Change in VRC07-523LS concentration among treated neonates and young infants | Measured through Week 24
  Based on laboratory evaluations
Presence of ARV genotypic resistance to drugs taken | Measured through Week 48
Presence of bNAb resistance as measured by inhibitory concentration | Measured through Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Chadwick, MD, Study Chair — Northwestern University Feinberg School of Medicine and Ann & Robert Lurie Children's Hospital of Chicago; Jennifer Jao, MD, Study Chair — Northwestern University Feinberg School of Medicine and Ann & Robert Lurie Children's Hospital of Chicago
Locations (50):
- United States (22):
  - 4601, University of California, San Diego Clinical Research Site, La Jolla, California
  - 5048, University of Southern California Clinical Research Site, Los Angeles, California
  - 5112, David Geffen School of Medicine at UCLA Clinical Research Site, Los Angeles, California
  - 5052, University of Colorado, Denver Clinical Research Site, Aurora, Colorado
  - 5055, South Florida CDTC Fort Lauderdale Clinical Research Site, Fort Lauderdale, Florida
  - 5051, University of Florida Center for HIV/AIDS Research, Education and Service (UF CARES) Clinical Research Site, Jacksonville, Florida
  - 5127, Pediatric Perinatal HIV Clinical Research Site, Miami, Florida
  - University of Miami CRS, Miami, Florida
  - Emory University School of Medicine NICHD CRS, Atlanta, Georgia
  - 5083, Rush University Cook County Hospital Clinical Research Site, Chicago, Illinois
  - 4001, Lurie Children's Hospital of Chicago Clinical Research Site, Chicago, Illinois
  - 5092, Johns Hopkins Clinical Research Site, Baltimore, Maryland
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - 5040, SUNY Stony Brook Clinical Research Site, Stony Brook, New York
  - 5114, Bronx Lebanon Hospital Center Clinical Research Site, The Bronx, New York
  - 5013, Jacobi Medical Center Clinical Research Site, The Bronx, New York
  - Philadelphia IMPAACT Unit CRS, Philadelphia, Pennsylvania
  - 6501, St Jude Children's Research Hospital Clinical Research Site, Memphis, Tennessee
  - Texas Children's Hospital CRS, Houston, Texas
  - 5128, Baylor College of Medicine/Texas Children's Hospital Clinical Research Site, Houston, Texas
  - Seattle Children's Research Institute CRS, Seattle, Washington
  - Univ. of Washington NICHD CRS, Seattle, Washington
- Hosp. General de Agudos Buenos Aires Argentina NICHD CRS, Buenos Aires, Argentina
- Brazil (6):
  - Hospital Nossa Senhora da Conceicao NICHD CRS, Porto Alegre, Rio Greande Do Sul
  - 5073, School of Medicine Federal University Minas Gerais Clinical Research Site, Minas Gerais
  - 5072, Hospital Federal dose Servidores do Estado Clinical Research Site, Rio de Janeiro
  - 5071, Instituto de Puericultura e Pediatria Martagao Gesteira Clinical Research Site, Rio de Janeiro
  - 5097, Hospital Geral de Nova Igaucu Clinical Research Site, Rio de Janeiro
  - 5074, University of Sao Paulo Clinical Research Site, São Paulo
- 30022, Les Centres GHESKIO Clinical Research Site, Port-au-Prince, Haiti
- 5121, Kenya Medical Research Institute/Walter Reed Project Clinical Research Center Kericho Clinical Research Site, Kericho, Kenya
- Malawi (2):
  - 12001, Malawi Clinical Research Site, Lilongwe, Central Region
  - 30301, Blantyre Clinical Research Site, Blantyre
- Puerto Rico (3):
  - 5129, University of Puerto Rico Gamma Project Clinical Research Site, San Juan, PR
  - University of Puerto Rico Pediatric HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan
- South Africa (4):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng
  - 30300, Umlazi Clinical Research Site, Durban, KwaZulu-Natal
  - 8950, FAMCRU Clinical Research Site, Tygerberg, Western Cape
- 5118, Kilimanjaro Christian Medical Centre Clinical Research Site, Moshi, Tanzania
- Thailand (2):
  - 5115, Siriraj Hospital Mahidol University Clinical Research Site, Bangkok, Bangkoknoi
  - 5116, Chiangrai Prachanukroh Hospital Clinical Research Site, Chiang Mai
- Uganda (3):
  - 31798, Baylor-Uganda Clinical Research Site, Kampala
  - MU-JHU Care Limited CRS, Kampala
  - MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala
- George CRS, Lusaka, Zambia
- Zimbabwe (3):
  - 30303, Saint Mary's Clinical Research Site, Chitungwiza
  - 30306, Seke North Clinical Research Site, Chitungwiza
  - 31890, Harare Family Care Clinical Research Site, Harare

REFERENCES:
- [Background] Persaud D, Bryson Y, Nelson BS, Tierney C, Cotton MF, Coletti A, Jao J, Spector SA, Mirochnick M, Capparelli EV, Costello D, Szewczyk J, Nicodimus N, Stranix-Chibanda L, Kekitiinwa AR, Korutaro V, Reding C, Carrington MN, Majji S, Yin DE, Jean-Philippe P, Chadwick EG. HIV-1 reservoir size after neonatal antiretroviral therapy and the potential to evaluate antiretroviral-therapy-free remission (IMPAACT P1115): a phase 1/2 proof-of-concept study. Lancet HIV. 2024 Jan;11(1):e20-e30. doi: 10.1016/S2352-3018(23)00236-9. Epub 2023 Dec 4. PMID 38061376
- [Background] Nelson BS, Tierney C, Persaud D, Jao J, Cotton MF, Bryson Y, Coletti A, Ruel TD, Spector SA, Reding C, Bacon K, Costello D, Perlowski C, Santos Cruz ML, Kosgei J, Majji S, Yin DE, Jean-Philippe P, Chadwick EG; IMPAACT P1115 Team. Infants Receiving Very Early Antiretroviral Therapy Have High CD4 Counts in the First Year of Life. Clin Infect Dis. 2023 Feb 8;76(3):e744-e747. doi: 10.1093/cid/ciac695. PMID 36031390
- [Background] Ruel TD, Capparelli EV, Tierney C, Nelson BS, Coletti A, Bryson Y, Cotton MF, Spector SA, Mirochnick M, LeBlanc R, Reding C, Zimmer B, Persaud D, Bwakura-Dangarembizi M, Naidoo KL, Hazra R, Jean-Philippe P, Chadwick EG. Pharmacokinetics and safety of early nevirapine-based antiretroviral therapy for neonates at high risk for perinatal HIV infection: a phase 1/2 proof of concept study. Lancet HIV. 2021 Mar;8(3):e149-e157. doi: 10.1016/S2352-3018(20)30274-5. Epub 2020 Nov 23. PMID 33242457
- [Derived] Persaud D, Coletti A, Nelson BS, Jao J, Capparelli EV, Costello D, Tierney C, Kekitiinwa AR, Nematadzira T, Njau BN, Moye J, Jean-Philippe P, Korutaro V, Nalugo A, Mbengeranwa T, Chidemo T, Mmbaga BT, Sakasaka PA, Cotton M, Jennings C, Hoffmann C, Hovind L, Bryson Y, Chadwick EG; IMPAACT P1115 Study Team. ART-free HIV-1 remission in children with in-utero HIV-1 after very early ART (IMPAACT P1115): a multicentre, open-label, phase 1/2 proof-of-concept study. Lancet HIV. 2025 Nov;12(11):e743-e752. doi: 10.1016/S2352-3018(25)00189-4. Epub 2025 Sep 25. PMID 41015049
- See also: Related Info — https://www.impaactnetwork.org/studies/p1115